CLINICAL TRIAL: NCT07169331
Title: A Phase 4, Single-Arm, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of Zanubrutinib in Chinese Patients With Treatment-Naive Waldenström Macroglobulinemia
Brief Title: A Study to Evaluate the Efficacy and Safety of Zanubrutinib in Chinese Adults With Treatment-Naive Waldenström Macroglobulinemia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-404
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Waldenström's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Participants will receive 160 mg zanubrutinib orally twice a day until progressive disease, unacceptable toxicity or death, withdrawal of consent, loss to follow-up, or study termination by the sponsor for any reason.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Administered orally
  Other Names: Brukinsa; BGB-3111

SUMMARY:
The purpose of this study is to measure the efficacy and safety with zanubrutinib in adults with Treatment-Naive (TN) Waldenström Macroglobulinemia (WM). The main objective of this Phase 4 study is to further characterize the efficacy of zanubrutinib in Chinese participants with TN WM in order to fulfill the post-marketing requirements from the National Medical Products Administration (NMPA). Safety data will be collected and evaluated in this study as well.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and definitive histologic diagnosis of WM. Participant must be treatment-naive.
* Participant must meet at least 1 criterion for treatment according to consensus panel criteria from the Seventh International Workshop on Waldenström's macroglobulinemia (IWWM).
* Participant must have measurable disease, as defined by serum immunoglobulin M (IgM) level > 0.5 g/dL.
* Participants must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* Participants must have adequate organ function as indicated by the following laboratory values ≤ 7 days before the first dose of study treatment:

  1. Participants must not have required blood transfusion or growth factor support ≤ 7 days before sample collection at screening for the following:

     * Absolute neutrophil count (ANC) ≥ 0.75 x 10^9/L.
     * Platelets ≥ 50 x 10^9/L.
  2. Creatinine clearance of ≥ 30 ml/min as estimated by the Cockcroft-Gault formula.
  3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN).
  4. Serum total bilirubin ≤ 2 x ULN (total bilirubin must be < 3 x ULN for participants with Gilbert syndrome).
* Female participants of childbearing potential must be willing to use a highly effective method of birth control and refrain from egg donation for the duration of the study and for at least 1 month after the last dose of zanubrutinib. They must also have a negative urine or serum pregnancy test result ≤ 7 days before the first dose of study treatment.

Exclusion Criteria:

* Evidence of disease transformation at the time of study entry.
* Central nervous system (CNS) involvement by WM. Patients with a history of CNS involvement must undergo magnetic resonance imaging (MRI) and cerebrospinal fluid cytology studies to document no evidence of CNS disease prior to study entry.
* Evidence of disease transformation at the time of study entry.
* Participants with any of the following cardiovascular risk factors:

  1. Active cardiac ischemia (eg, cardiac chest pain) ≤ 28 days before first dose of study drug.
  2. Any history of acute myocardial infarction ≤ 6 months before the first dose of study drug.
  3. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV (Appendix 7)≤ 6 months before the first dose of study drug.
  4. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before the first dose of study drug.
  5. Active, clinically significant second-degree atrioventricular block Mobitz II, or third degree atrioventricular block.
  6. Any history of cerebrovascular accident ≤ 6 months before the first dose of study drug.
  7. Uncontrolled hypertension that cannot be managed by standard antihypertension medications ≤ 28 days before the first dose of study drug.
  8. Any episode of syncope or seizure ≤ 28 days before first dose of study drug.
* At the time of study entry, participants taking warfarin or other vitamin K antagonists.
* Participants requiring ongoing therapy with strong or moderate cytochrome CYP3A inducers
* Corticosteroids given with antineoplastic intent within 7 days, or chemotherapy, targeted therapy, or radiation therapy within 4 weeks, or antibody-based therapy within 4 weeks before the start of study drug.
* Major surgical procedure within 4 weeks before the start of study treatment (bone marrow aspirate and biopsy procedures are not considered major surgical procedures).

Note: Other protocol defined criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Complete Response (CR) or Very Good Partial Response (VGPR) as Assessed by the Investigator | Up to approximately 33 Months
  The percentage of participants who achieve either a complete response or very good partial response (VGPR) as determined by the investigator using an adaptation of the response criteria updated at the Sixth International Workshop on Waldenström's macroglobulinemia (IWWM).

SECONDARY OUTCOMES:
Major Response Rate (MRR) as Assessed by the Investigator | Up to approximately 33 Months
  MRR is defined as the percentage of participants achieving CR, VGPR, or partial response (PR) as determined by the investigator per the modified IWWM criteria.
Duration of Major Response (DOMR) as Assessed by the Investigator | Up to approximately 33 Months
  DOMR is defined as the time from first determination of response (CR, VGPR, or PR) (per modified IWWM criteria) until first documentation of disease progression (per modified IWWM criteria) or death, whichever comes first
Progression-free Survival (PFS) as Assessed by the Investigator | Up to approximately 33 Months
  Progression-free survival (PFS) as assessed by the investigator, defined as time from start of treatment to the first documentation of disease progression (per modified IWWM criteria) or death, whichever occurs first.
Number of Participant with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose of study drug until 30 days after the last dose, up to approximately 33 months
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory values, vital signs, physical examination findings, and electrocardiogram results.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (8):
- China (8):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central Peoples Hospital, Yichang, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/